CLINICAL TRIAL: NCT02298777
Title: Metabolomic Analysis of Systemic Sclerosis
Acronym: SCLEROMICS
Status: Terminated | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5723
Record Dates: First submitted 2014-11-06; First posted 2014-11-24 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Scleroderma (Limited and Diffuse); Undifferentiated Connective Tissue Disease; Raynaud Disease; Vascular Disease; Healthy Control Subjects
MeSH Terms: conditions — Scleroderma, Diffuse; Undifferentiated Connective Tissue Diseases; Raynaud Disease; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Scleroderma (SSc) patients (beginners and established forms).: Patients with the ACR / EULAR (2012) and / or criteria of Leroy and Medsger (2001)
  Biological samples (skin, urine and blood):
  * 1st point at patient's inclusion visit
  * 2nd point (optional) at SSc patient's visceral complication (assessed during 3 years)
  Interventions: Procedure: - Skin biopsy - Urine sample - Blood sample
- Undifferentiated Connective Tissue Disease (UCDT) patients: Patients with criteria proposed by Mosca et al. (1998)
  Biological samples (skin, urine and blood):
  - 1single point at patient's inclusion visit
  Interventions: Procedure: - Skin biopsy - Urine sample - Blood sample
- Raynaud disease patients: Patients with primary and isolated Raynaud disease
  Biological samples (skin, urine and blood):
  - 1single point at patient's inclusion visit
  Interventions: Procedure: - Skin biopsy - Urine sample - Blood sample
- Vascular disease patients: Patients with vascular disease (type 2 diabetes, occlusive vascular disease, history of myocardial infarction or ischemic stroke)
  Biological samples (skin, urine and blood):
  - 1single point at patient's inclusion visit
  Interventions: Procedure: - Skin biopsy - Urine sample - Blood sample
- Healthy control subjects: Healthy subjects (no sign of connective tissue disease, no Raynaud, no vascular disease)
  Biological samples (skin, urine and blood):
  - 1single point at patient's inclusion visit
  Interventions: Procedure: - Skin biopsy - Urine sample - Blood sample

INTERVENTIONS:
Procedure: - Skin biopsy - Urine sample - Blood sample

SUMMARY:
Currently investigators do not have diagnostic and prognostic markers for SSc which almost always starts with a vascular disease (Raynaud's disease) isolated for several years.

The primary purpose is to highlight discriminating metabolic profiles depending on the characteristics of the disease, allowing early diagnosis of SSc at the onset of vascular lesions, by comparing the profiles of SSc beginners (<3 years) to established forms (> 3 years).

Secondary purposes:

* Prognosis: to study the metabolomics profile of SSc when a visceral complication occurs
* Diagnosis: to compare the metabolomics profile of SSc to undifferentiated connective tissue disease (UCDT), Raynaud's disease (RD), vascular disease (VD) and healthy controls
* Exploratory: to compare the metabolomics profile of blood, urine and skin of SSc patients

ELIGIBILITY:
Inclusion criteria:

* Group 1 (scleroderma) : Patients with ACR / EULAR (2012) and / or criteria of Leroy and Medsger (2001)
* Group 2 (UCDT) : Patients with criteria proposed by Mosca et al. (1998)
* Group 3 (Raynaud) : Patients with primary and isolated Raynaud disease
* Group 4 (vascular disease) : Patients with type 2 diabetes, occlusive vascular disease, history of myocardial infarction or ischemic stroke
* Group 5 (healthy control) : healthy subjects (no sign of connective tissue disease, no Raynaud, no vascular disease)

Exclusion criteria:

* Group 1 (scleroderma) : Patients not fulfilling ACR / EULAR (2012) and / or criteria of Leroy and Medsger (2001), or with another auto-immune disease
* Group 2 (UCDT) : Patients not fulfilling criteria proposed by Mosca et al. (1998)
* Group 3 (Raynaud) : Patients with no Raynaud disease
* Group 4 (vascular disease) : Patients with no vascular disease
* Group 5 (healthy control) : Patients with sign of connective tissue disease, Raynaud, or vascular disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with systemic sclerosis (SSc),
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
change of metabolomics profiles between SSc beginners (<3 years) and SSc established forms (> 3 years) at baseline inclusion. | 1 point at patient's inclusion visit
  Metabolomic profiles will be classified in a database and compared.

SECONDARY OUTCOMES:
Study and comparison of discriminating metabolomics profiles for prognosis, diagnosis and exploration of SSc. | 1st point at patient's inclusion visit (all arms) + 2nd point at patient's complication (group1) during 3 years
  Metabolomic profiles will be classified in a database and compared between each other's (SSc, UCDT, RD, VD and healthy control arms) We will look for a correlation between these profiles and the evolution of clinical and biological characteristics of SSc (SSc arm)

CONTACTS AND LOCATIONS:
Overall Officials: Chatelus Emmanuel, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (4):
- France (4):
  - CHU, Dijon
  - Hôpitaux privés de Metz, Metz
  - CHU, Reims
  - Hôpitaux Universitaires de Strasbourg, Strasbourg